CLINICAL TRIAL: NCT02022657
Title: PrEP Adherence Monitoring Using Dried Blood Spots
Brief Title: Pre-Exposure Prophylaxis (PrEP) Adherence Monitoring Using Dried Blood Spots
Acronym: DOT-DBS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: San Francisco Department of Public Health (Other Government); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 13-0427; U01AI106499 (NIH)
Record Dates: First submitted 2013-12-09; First posted 2013-12-30 (Estimated); Results first posted 2019-04-18 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: PrEP Adherence Monitoring
Keywords: Pre exposure prophylaxis; Dried blood spots
MeSH Terms: interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Tenofovir; Emtricitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 33%/67% (Active Comparator): Participants will be randomized to one of 6 sequences consisting of two directly observed dosing regimens expressed as % of daily dosing of Truvada
  Interventions: Drug: Truvada
- 33%/100% (Active Comparator): Participants will be randomized to one of 6 sequences consisting of two directly observed dosing regimens expressed as % of daily dosing of Truvada
  Interventions: Drug: Truvada
- 67%/33% (Active Comparator): Participants will be randomized to one of 6 sequences consisting of two directly observed dosing regimens expressed as % of daily dosing of Truvada
  Interventions: Drug: Truvada
- 67%/100% (Active Comparator): Participants will be randomized to one of 6 sequences consisting of two directly observed dosing regimens expressed as % of daily dosing of Truvada
  Interventions: Drug: Truvada
- 100%/33% (Active Comparator): Participants will be randomized to one of 6 sequences consisting of two directly observed dosing regimens expressed as % of daily dosing of Truvada
  Interventions: Drug: Truvada
- 100%/67% (Active Comparator): Participants will be randomized to one of 6 sequences consisting of two directly observed dosing regimens expressed as % of daily dosing of Truvada
  Interventions: Drug: Truvada

INTERVENTIONS:
Drug: Truvada — Truvada is a combination pill consisting of tenofovir and emtricitabine used in PrEP
  Other Names: Tenofovir; Emtricitabine

SUMMARY:
The primary objective of this study is to define the mean, variance, and dose proportionality for tenofovir-diphosphate(TFV-DP) in dried blood spots resulting from 33%, 67%, and 100% of daily dosing with 200mg emtricitabine and 300mg of tenofovir disoproxil fumarate (as Truvada®). With this information, a model will be established to predict adherence rates to TFV-DP using DBS. Forty-eight healthy HIV-uninfected adult participants who are at low risk for HIV infection will be randomized to one of 6 sequences consisting of two directly observed dosing regimens, 33%/67%, 33%/100%, 67%/33%, 67%/100%, 100%/33%, and 100%/67% with each dose regimen lasting approximately 12 weeks, separated by an approximately 12 week washout period. DBS will be collected at regular intervals, including during the washout. The hypothesis of the study is that levels of TFV-DP in DBS will predict adherence rates in the preceding 1-3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Ambulatory 18-50 year old adults. Enrollment will target approximately half women and approximately one third African-Americans and one third Latino.
2. Ability to comply with study procedures, including directly observed dosing visits and availability and use of audio-video streaming technology.

Exclusion Criteria:

1. Inability to give informed consent
2. A minimum scalp hair length of 2 cm in the occipital region.
3. Pregnancy or plan to become pregnant or unwillingness to use birth control
4. Current breastfeeding.
5. High risk of HIV-1 infection (for example: sexually active with an HIV infected partner; men who have sex with men who may engage in condom-less intercourse with HIV-infected partners or partner of unknown status during the study; males or females who exchange sex for money, shelter, or gifts; active injection drug use or during the last 12 months; newly diagnosed sexually transmitted infections in last 6 months)
6. Positive screening HIV+ ELISA or suspected acute HIV infection in the opinion of the clinician. (example signs and symptoms of acute HIV infection include combinations of fever, headache, fatigue, arthralgia, vomiting, myalgia, diarrhea, pharyngitis, rash, night sweats, and adenopathy cervical or inguinal)
7. Positive Hepatitis B (HBV) surface antigen test at screening
8. Active psychiatric illness, social condition, or alcohol/drug abuse that, in the opinion of the investigators, would interfere with study requirements.
9. History of non-traumatic, pathologic bone fractures
10. Glomerular Filtration Rate (GFR, creatinine clearance) < 60 ml/min (MDRD equation).
11. Urine dipstick protein ≥ 2+
12. Total bilirubin and/or hepatic transaminases (ALT and AST) ≥ 2.5x upper limit of normal
13. Absolute neutrophil count ≤ 1,500/mm3, platelets count ≤ 100,000/mm3, or hemoglobin ≤ 10 g/dL.
14. Medical condition that alters red blood cell kinetics including hemoglobinopathies or active hemolysis.
15. Any laboratory value or uncontrolled medical conditions that would interfere with the study conditions such as, heart disease and/or cancer.
16. Contraindicated concomitant medications (including investigational agents, aminoglycosides, ganciclovir/valganciclovir, chronic high-dose acyclovir/valacyclovir, cyclosporine, amphotericin B, foscarnet, and cidofovir, and products with same or similar active ingredients as the study medications (Truvada®) including ATRIPLA®, COMPLERA®, EMTRIVA®, VIREAD®; or drugs containing lamivudine or adefovir, which are close analogs of Emtricitabine (FTC) and tenofovir, respectively).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter L Anderson, PharmD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of California San Francisco/San Francisco Department of Public Health, San Francisco, California
  - University of Colorado Denver, Aurora, Colorado

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD

REFERENCES:
- [Background] Anderson PL, Liu AY, Castillo-Mancilla JR, Gardner EM, Seifert SM, McHugh C, Wagner T, Campbell K, Morrow M, Ibrahim M, Buchbinder S, Bushman LR, Kiser JJ, MaWhinney S. Intracellular Tenofovir-Diphosphate and Emtricitabine-Triphosphate in Dried Blood Spots following Directly Observed Therapy. Antimicrob Agents Chemother. 2017 Dec 21;62(1):e01710-17. doi: 10.1128/AAC.01710-17. Print 2018 Jan. PMID 29038282
- [Derived] Ibrahim ME, Castillo-Mancilla JR, Yager J, Brooks KM, Bushman L, Saba L, Kiser JJ, MaWhinney S, Anderson PL. Individualized Adherence Benchmarks for HIV Pre-Exposure Prophylaxis. AIDS Res Hum Retroviruses. 2021 Jun;37(6):421-428. doi: 10.1089/AID.2020.0108. Epub 2020 Dec 10. PMID 33191774
- [Derived] Grant RM, Pellegrini M, Defechereux PA, Anderson PL, Yu M, Glidden DV, O'Neal J, Yager J, Bhasin S, Sevelius J, Deutsch MB. Sex Hormone Therapy and Tenofovir Diphosphate Concentration in Dried Blood Spots: Primary Results of the Interactions Between Antiretrovirals And Transgender Hormones Study. Clin Infect Dis. 2021 Oct 5;73(7):e2117-e2123. doi: 10.1093/cid/ciaa1160. PMID 32766890
- [Derived] Koss CA, Liu AY, Castillo-Mancilla J, Bacchetti P, McHugh C, Kuncze K, Morrow M, Louie A, Seifert S, Okochi H, MaWhinney S, Gandhi M, Anderson PL. Similar tenofovir hair concentrations in men and women after directly observed dosing of tenofovir disoproxil fumarate/emtricitabine: implications for preexposure prophylaxis adherence monitoring. AIDS. 2018 Sep 24;32(15):2189-2194. doi: 10.1097/QAD.0000000000001935. PMID 30212404
- [Derived] Castillo-Mancilla J, Seifert S, Campbell K, Coleman S, McAllister K, Zheng JH, Gardner EM, Liu A, Glidden DV, Grant R, Hosek S, Wilson CM, Bushman LR, MaWhinney S, Anderson PL. Emtricitabine-Triphosphate in Dried Blood Spots as a Marker of Recent Dosing. Antimicrob Agents Chemother. 2016 Oct 21;60(11):6692-6697. doi: 10.1128/AAC.01017-16. Print 2016 Nov. PMID 27572401

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 52 subjects from 2 sites were analyzed-- CU enrolled only 34.
Groups:
- 100% First, Then 67%: 100% dosing: Dose every day for ~12 weeks 67% holiday dosing regimen: 2 weeks on medication, 1 week off, repeat for ~ 12 weeks 67% intermittent dosing regimen: 2 days on medication, 1 day off, repeat for ~ 12 weeks
  67% Intermittent and 67% Holiday dosing combined for analysis.
- 100% First, Then 33%: 100% dosing regimen: dosing every day for ~12 weeks 33% holiday dosing regimen: 1 week on medication, 2 weeks off, repeat for ~ 12 weeks 33% intermittent dosing regimen:1 day on medication, 2 days off, repeat for ~ 12 weeks
  33% Intermittent and 33% Holiday dosing combined for analysis.
- 67% First, Then 100%: 67% holiday dosing regimen: 2 weeks on medication, 1 week off, repeat for ~ 12 weeks 67% intermittent dosing regimen: 2 days on medication, 1 day off, repeat for ~ 12 weeks 100% dosing regimen: dosing every day, repeat for ~12 weeks
  67% Intermittent and 67% Holiday dosing combined for analysis.
- 67% First, Then 33%: 67% holiday dosing regimen: 2 weeks on medication, 1 week off, repeat for ~ 12 weeks 67% intermittent dosing regimen: 2 days on medication, 1 day off, repeat for ~ 12 weeks 33% holiday dosing regimen: 1 week on medication, 2 weeks off, repeat for ~ 12 weeks 33% intermittent dosing regimen:1 day on medication, 2 days off, repeat for ~ 12 weeks
  67% Intermittent and 67% Holiday dosing combined for analysis. 33% Intermittent and 33% Holiday dosing combined for analysis.
- 33% First, Then 100%: 33% holiday dosing regimen: 1 week on medication, 2 weeks off, repeat for ~ 12 weeks 33% intermittent dosing regimen:1 day on medication, 2 days off, repeat for ~ 12 weeks 100% dosing: Dose every day for ~12 weeks
  33% Intermittent and 33% Holiday dosing combined for analysis.
- 33% First, Then 67%: 33% holiday dosing regimen: 1 week on medication, 2 weeks off, repeat for ~ 12 weeks 33% intermittent dosing regimen:1 day on medication, 2 days off, repeat for ~ 12 weeks 67% holiday dosing regimen: 2 weeks on medication, 1 week off, repeat for ~ 12 weeks 67% intermittent dosing regimen: 2 days on medication, 1 day off, repeat for ~ 12 weeks
  33% Intermittent and 33% Holiday dosing combined for analysis. 67% Intermittent and 67% Holiday dosing combined for analysis.
Period: Overall Study
Arm/Group | 100% First, Then 67% | 100% First, Then 33% | 67% First, Then 100% | 67% First, Then 33% | 33% First, Then 100% | 33% First, Then 67%
Started | 10 | 8 | 9 | 8 | 8 | 9
Completed | 8 | 8 | 8 | 8 | 8 | 8
Not Completed | 2 | 0 | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Arms were combined to be consistent with protocol subject randomization. Subjects were randomized to one of six arms. "Holiday" and "intermittent" groups for 33 and 67% dosing were combined because drug concentrations didn't differ between groups (PMID: 29038282). Combined arms best categorize the study and population.
Groups:
- All Dosing Regimens: Baseline characteristics for all 48 subjects included in analysis. Baseline characteristics not stratified based on dosing regimen.
Arm/Group | All Dosing Regimens
Number analyzed (Participants) | 48
Age, Continuous [Median (Full Range); unit: years] | 29 [21 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 26
  Hispanic | 14
  Black/African American | 8

OUTCOME MEASURES:

1. Primary Outcome: Steady State Concentrations of TFV-DP for Different Dosing Patterns of Truvada
Description: TFV-DP concentrations in DBS respective to dosing regimens of 33%, 67%, 100% of daily dosing.
Time Frame: Assessed every 2 weeks during the dosing periods and at steady-state, week 12 for the first dosing period and week 36 for the second dosing period.
Population: The total number of participants was 48. Each participant was randomized to 2 of 3 dosing regimens for a total of 32 participants each, however 2 participants completed only the first regimen.
Measure: Mean (Standard Deviation); unit: fmol/punch
Groups:
- DOT-DBS Dosing 33%: 33%
- DOT-DBS Dosing 67%: 67%
Arm/Group | DOT-DBS Dosing 33% | DOT-DBS Dosing 67% | DOT-DBS Dosing 100%
Number analyzed (Participants) | 30 | 32 | 32
fmol/punch | 530 (159) | 997 (267) | 1605 (405)

ADVERSE EVENTS:
Time Frame: Time of consenting to study exit (Week 36 or earlier), Max 10 months.
Description: AEs were graded per the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, V1.0 Aug 2009 (US Dept HHS, NIH, NIAID) Available from: http://rsc.tech-res.com/docs/default-source/safety/table_for_grading_severity_of_adult_pediatric_adverse_events.pdf
  Arms were combined as Truvada was FDA approved for daily use (100% dosing) at the time of study initiation- no arm was considered to be more at risk for AEs than another.
Groups:
- All Dosing Regimens: Overall, the study showed an unremarkable and expected AE profile. At study initiation Truvada was FDA approved for daily dosing (100% daily dosing). Thus, the AE profile was already established for 100% dosing and AE rates in the lower doses (33% and 67%) would not exceed the established rate for daily dosing (100%). This study was not designed to collect new safety data or to update the established AE/Safety profiles for Truvada. Therefore AE data was combined for all dosing regimens since AEs reported per arm/group are not meaningful for research or clinical applications.
Arm/Group | All Dosing Regimens
All-Cause Mortality (participants affected / at risk) | 0/48
Serious Adverse Events (participants affected / at risk) | 1/48
Other Adverse Events (participants affected / at risk) | 48/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Dosing Regimens (N=48)
Anxiety (Psychiatric disorders) | 1 (1) — Not related to study medication; anxiety requiring hospitalization and medication
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Dosing Regimens (N=48)
Cold Symptoms (General disorders) | 41 (83)
Abdominal Pain (Gastrointestinal disorders) | 14 (17)
Diarrhea (Gastrointestinal disorders) | 7 (12)
Headache (General disorders) | 7 (10)
Nausea (Gastrointestinal disorders) | 15 (24)
Vomitting (Gastrointestinal disorders) | 4 (7)
Fatigue (General disorders) | 14 (16)
Loss of Appetite (General disorders) | 3 (5)
Abnormal Labs (General disorders) | 32 (88) — Lab, # of Incidents ALT, 5 AST, 4 Bilirubin, 9 Calcium, 2 Glucose, 16 Hg, 2 Lipase, 4 Other, 7 Phosphorous, 24 Potassium, 3 RBC, 1 Sodium, 1 UA- Protein, 6 UA-RBC, 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No